CLINICAL TRIAL: NCT02049073
Title: Zonisamide and Methylprednisolone to Prevent Noise-induced Temporary Hearing Loss
Brief Title: Prevention of Noise-induced Hearing Loss
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: new data makes this trial unethical
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Judith Lieu, Associate Professor of Otolaryngology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIHL2014
Record Dates: First submitted 2014-01-23; First posted 2014-01-29 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Noise-induced Hearing Loss
Keywords: hearing loss; noise induced hearing loss; zonisamide
MeSH Terms: conditions — Hearing Loss, Noise-Induced; Hearing Loss | interventions — Zonisamide; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Zonisamide (Experimental): Zonisamide 100 mg or 200 mg pill administered orally every day for 2 weeks
  Interventions: Drug: Zonisamide
- Methylprednisolone (Experimental): Methylprednisolone 32 mg or 64 mg pill administered orally once
  Interventions: Drug: Methylprednisolone
- Control (No Intervention): no medication

INTERVENTIONS:
Drug: Zonisamide — Zonisamide 100 mg or 200 mg pill administered orally every day for 2 weeks
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Methylprednisolone — Methylprednisolone 32 mg or 64 mg pill administered orally once
  Other Names: Medrol; Solu-Medrol; Depo-Medrol; Hybrisil; A-Methapred
  Arms: Methylprednisolone

SUMMARY:
Noise-induced hearing loss affects an estimated 5% of the worldwide population, with 30-40 million Americans exposed to hazardous sound or noise levels regularly. Sources of noise may be occupational, blast noise, or recreational. Trauma to the inner ear can occur through transient hearing loss or permanent hearing loss. Although hearing recovers after temporary transient hearing loss, growing evidence suggests that repeated temporary transient hearing loss may lead to a permanent hearing loss. Currently, there are no treatments and there are no known medications that can be used clinically to prevent noise-induced hearing loss in humans.

The long-term goal of this research is to find medications that can prevent noise-induced hearing loss. The purpose of the present pilot study is to evaluate zonisamide and methylprednisolone as medications to prevent temporary transient hearing loss in humans.

DETAILED DESCRIPTION:
Noise-induced hearing loss (NIHL) affects an estimated 5% of the worldwide population, with 30-40 million Americans exposed to hazardous sound or noise levels regularly. Sources of noise may be occupational (e.g., manufacturing, construction), blast noise (e.g., firearms or explosions), or recreational (e.g., loud music, power tools). Trauma to the inner ear can occur through transient hearing loss (temporary threshold shifts, TTS) or permanent hearing loss (permanent threshold shift, PTS). Although hearing recovers after a TTS in about 24-48 hours, growing evidence suggests that repeated TTS may lead to PTS. Both TTS and PTS lead to a decrease in hearing thresholds at 3000 to 6000 Hz.

Currently, there are no treatments for human NIHL although this is an area of active investigation. Protection against NIHL consists of limiting noise exposure through Occupational Safety and Health Administration (OSHA) limits to occupational noise and the wearing of hearing-protection devices (e.g., ear muffs or earplugs). There are no known medications that can be used clinically to prevent NIHL in humans.

LePrell and colleagues have successfully established a protocol for inducing TTS using digitally-modified pop or rock music. This model of experimentally-induced TTS was intended to provide an ethical way of testing medications that might prevent NIHL.

In a mouse model, Bao and colleagues were able to use zonisamide, an anti-epileptic medication approved for the treatment of partial seizures, and methylprednisolone, a glucocorticoid medication, to protect against noise-induced PTS. The long-term goal of this research is to find medications that can prevent NIHL. The goal of the present pilot study is to evaluate zonisamide and methylprednisolone as medications to prevent TTS in humans.

Specific Aim 1: Examine zonisamide as a possible prophylactic medication to prevent noise-induced hearing loss, using an escalating dose protocol. Healthy volunteers would be given 100 or 200 mg of zonisamide as one-time doses or as a daily medication for two week (to establish a steady-state). They would be exposed to digitally-modified pop or rock music for 4 hours and undergo serial testing of hearing and monitoring for side effects after their sound exposure for 3-4 hours. They would be monitored at one day and one week post-exposure for hearing and other side effects.

Hypothesis: Zonisamide is able to protect against noise-induced hearing loss in humans.

Specific Aim 2: Examine methylprednisolone as a possible prophylactic medication to prevent noise-induced hearing loss, using an escalating dose protocol. Healthy volunteers would be given 32 or 64 mg of methylprednisolone as one-time doses. They would undergo the same music exposure and post-sound exposure monitoring as described above.

Hypothesis: Methylprednisolone is able to protect against noise-induced hearing loss in humans

ELIGIBILITY:
Inclusion Criteria:

* adults 18 to 30 years old
* normal hearing
* good to excellent health

Exclusion Criteria:

* hearing loss
* history of seizures
* history of allergy or hypersensitivity to sulfonamide or oral steroid medications

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Pure Tone Thresholds | 15 minutes post-music exposure
  The primary outcome will be pure tone hearing thresholds (particularly 2000, 3000, 4000, and 6000 Hz) as measured by audiogram in a soundproof booth.

SECONDARY OUTCOMES:
DPOAE | visit 2, pre-music exposure; visit 3-one week after music exposure
  Distortion-product otoacoustic emissions (DPOAE) will be used as a secondary auditory outcome. A tinnitus questionnaire (Tinnitus Handicap Inventory) will be used to measure the secondary outcome of tinnitus, which frequently accompanies TTS.
Pure tone thresholds | 1 hr 15 min, 2 hr 15 min, and 3 hr 15 min post exposure.
  This outcome measures recovery of hearing after loud music exposure

OTHER OUTCOMES:
Pure tone thresholds | One week after music exposure.
  Recovery of hearing after noise exposure

CONTACTS AND LOCATIONS:
Overall Officials: Judith Lieu, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
undecided